CLINICAL TRIAL: NCT00633659
Title: A Phase II Study of Hemospan® Versus Voluven® to Evaluate Vascular Resistance and Forearm Blood Flow, and to Assess Local Skin Blood Flow and Tissue Oxygenation in the Ischemic Foot of Patients With Chronic Critical Limb Ischemia
Brief Title: Pilot Study of Hemospan® in Patients With Chronic Critical Limb Ischemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sangart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 6034
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Vascular Disease; Critical Lower Limb Ischemia
Keywords: Hemospan; Oxygen carriers; Blood substitutes; Ischemia; Tissue oxygenation
MeSH Terms: conditions — Vascular Diseases; Ischemia | interventions — maleimide-polyethylene glycol-modified hemoglobin, MP4; HES 130-0.4; Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemospan (MP4OX) (Experimental): 4.3 g/dL MalPEG-Hb solution
  Interventions: Drug: Hemospan (MP4OX)
- Control (Experimental): Voluven (HES 130/0.4)
  Interventions: Drug: Voluven (HES 130/0.4)

INTERVENTIONS:
Drug: Hemospan (MP4OX) — 250 mL of Hemospan (MP4OX)
  Other Names: MP4OX solution; 4.3 g/dL MalPEG-Hb; PEGylated Hb
  Arms: Hemospan (MP4OX)
Drug: Voluven (HES 130/0.4) — 250 mL of Voluven (HES 130/0.4) solution
  Other Names: 6% hetastarch solution; 6% HES 130/0.4
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effects of Hemospan infusion on vascular reactivity, regional perfusion and oxygenation of ischemic tissue in patients with chronic critical lower limb ischemia.

DETAILED DESCRIPTION:
Hemospan® is a novel hemoglobin-based oxygen carrier developed to perfuse and oxygenate tissue at risk for ischemia and hypoxia. Because of its molecular size and oxygen binding characteristics, Hemospan selectively off-loads oxygen in tissues predisposed to low oxygen tension. Preclinical evidence suggests that Hemospan provides volume expansion and enhances tissue perfusion. Hemospan is therefore being developed as an oxygen-carrying plasma expander for patients where tissues are at risk of inadequate perfusion and oxygenation.

In patients with chronic critical lower limb ischemia (CCLI), the primary cause of ischemic symptoms in the leg is insufficient perfusion. As many of the patients suffering from CCLI are elderly and have concomitant disease, surgical procedures may not always be possible. The goal of all treatments is to improve the blood flow in the nutritional vessels of the ischemic areas; one such possibility may be to use an oxygen-carrying plasma expander.

Hemospan has been shown to improve the oxygenation of tissues by preserving functional capillary density. In addition, Hemospan has a high affinity for oxygen - a feature that is specifically designed to target the unloading of oxygen in the microcirculation where local PO2 levels are much lower (e.g., in ischemic regions). Since Hemospan is a cell-free oxygen carrier, it should be able to perfuse capillaries that are so constricted that red blood cells are unable to flow through them.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female (surgically sterile or post-menopausal) patients with CCLI that meet the following definition: i) History of pain at rest and/or ulceration; ii) Ankle systolic BP/Brachial systolic BP Index (ABI) <0.6 at the time of inclusion; iii) Ankle systolic BP <70 mmHg and/or toe systolic BP <50 mmHg
* Has received written and verbal information about the investigational product and the protocol by the investigator and has had the opportunity to ask questions about the study
* Patients must sign an Informed Consent Form (ICF), that has been reviewed and approved by the independent Ethics Committee (EC)

Exclusion Criteria:

* Severe congestive heart failure (EF <40%, or New York Heart Association Class III or IV
* Any acute or chronic condition that will limit the patient's ability to complete the study
* Recent acute coronary syndrome (unstable angina or myocardial infarction [MI] within 1 month)
* Severe dementia or clinically significant psychiatric disorder requiring active treatment
* Evidence of untreated or uncontrolled hypertension (SBP >180 mmHg, or DBP >100 mmHg), or a difference in systolic BP in each arm that is >15 mmHg (measured by cuff and a pen-Doppler at screening in the supine position, in both arms)
* Smoking or use of any nicotine-containing product (e.g., snuff) within previous 24 hours before start of study
* Any systemic rheumatic disease
* Taking oral steroid therapy (does not include steroids taken intermittently via inhaler)
* Chronic hepatic disease (abnormal LFTs >3X upper limit of normal, known history of Hepatitis C or B)
* Chronic renal disease (creatinine >1.8 mg/dL, or known polycystic kidney disease)
* Expectation of poor patient compliance with study protocol
* Patients scheduled for surgical procedure within 7 days from start of this study
* Involved in any investigational drug or device trial within 30 days prior to this study
* Professional or ancillary personnel involved with this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of Hemospan on vascular resistance by evaluating blood flow in the forearm | 4 hours

SECONDARY OUTCOMES:
To evaluate the effects of Hemospan on local skin blood flow and tissue oxygenation in an ischemic region of the foot | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pär Olofsson, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska Universitetssjukhuset, Stockholm, Sweden

REFERENCES:
- [Background] Bjorkholm M, Fagrell B, Przybelski R, Winslow N, Young M, Winslow RM. A phase I single blind clinical trial of a new oxygen transport agent (MP4), human hemoglobin modified with maleimide-activated polyethylene glycol. Haematologica. 2005 Apr;90(4):505-15. PMID 15820947
- [Background] Olofsson C, Ahl T, Johansson T, Larsson S, Nellgard P, Ponzer S, Fagrell B, Przybelski R, Keipert P, Winslow N, Winslow RM. A multicenter clinical study of the safety and activity of maleimide-polyethylene glycol-modified Hemoglobin (Hemospan) in patients undergoing major orthopedic surgery. Anesthesiology. 2006 Dec;105(6):1153-63. doi: 10.1097/00000542-200612000-00015. PMID 17122578
- [Background] Olofsson C, Nygards EB, Ponzer S, Fagrell B, Przybelski R, Keipert PE, Winslow N, Winslow RM. A randomized, single-blind, increasing dose safety trial of an oxygen-carrying plasma expander (Hemospan) administered to orthopaedic surgery patients with spinal anaesthesia. Transfus Med. 2008 Feb;18(1):28-39. doi: 10.1111/j.1365-3148.2007.00811.x. PMID 18279190
- [Background] Winslow RM. Red cell substitutes. Semin Hematol. 2007 Jan;44(1):51-9. doi: 10.1053/j.seminhematol.2006.09.013. PMID 17198847
- See also: For more information about Sangart, Inc. — http://sangart.com